CLINICAL TRIAL: NCT04660110
Title: Evaluation of the Household-level Impact of a Single Round of Intermittent Preventive Treatment of Malaria in Schoolchildren: A Randomized Study
Brief Title: Household-level Impact of IPT of Malaria in Schoolchildren
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Lecturer, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SBMC_HH impact
Record Dates: First submitted 2020-11-09; First posted 2020-12-09 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — adenylate isopentenyltransferase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): A single dose/round of IPT with DP (40mg/320mg tabs, Fosun Pharmaceuticals)
  Interventions: Drug: IPT with Dihydroartemisinin Piperaquine
- Standard of care (No Intervention): Health information, no study drugs

INTERVENTIONS:
Drug: IPT with Dihydroartemisinin Piperaquine — A single dose/round of IPT with Dihydroartemisinin Piperaquine (40mg/320mg tabs, Fosun Pharmaceuticals)
  Arms: Intervention arm

SUMMARY:
The study will evaluate the household-level impact of IPT for malaria in schoolchildren on malaria transmission, using a randomized trial design. Two schools in Busia district will be randomly selected and randomize to either IPT with dihydroartemisinin piperaquine (DP, IPT arm), or standard of care (no intervention). A single dose/round of IPT with DP (40mg/320mg tabs, Fosun Pharmaceuticals) will be given to the children in the intervention arm. The full dose will be given as oral tablets once a day for 3 consecutive days to all eligible children in the intervention school. Surveys will be conducted in households of 100 randomly selected children in each of the study arms at baseline, one month and three months following the intervention. The target population will include all household members of the selected households.

DETAILED DESCRIPTION:
The most promising strategy to address the burden of malaria in school-aged children is intermittent preventive treatment with antimalarials (IPTsc). IPTsc has clearly been demonstrated to improve the health and educational attainment of schoolchildren. While the goal of IPTsc is improving the individual outcomes, reducing infections in schoolchildren, a primary reservoir for human-to-mosquito transmission may reduce overall transmission increasing the benefits and adding value to this intervention. In areas where the burden of malaria remains high despite implementation of currently available tools, IPTsc could act as a complimentary measure to reduce transmission incrementally while decreasing the burden of malaria in a vulnerable, high yield population. However, the benefits of IPTsc specifically targeting transmission reduction, have not widely been evaluated. We will evaluate impact of IPTsc with an antimalarial in schoolchildren on the malaria burden in household members in a high transmission area. The objective is to:

1. To determine the impact of intermittent preventive treatment of malaria in schoolchildren on malaria transmission at the household, as measured by the prevalence of parasitaemia at the household level.
2. To determine the impact of intermittent preventive treatment of malaria in schoolchildren on the health of the children as measured by the prevalence of parasitaemia among the children.

Two primary schools will be randomly selected from the list of the schools in Busia district. The list will act as the sampling frame for the school selection. Following the identification of the two schools to participate in the study. The schools will be randomized to either intervention or control arm.

A single dose/round of IPT with DP (40mg/320mg tabs, Fosun Pharmaceuticals) will be given to the children in the intervention arm. The full dose will be given as oral tablets once a day for 3 consecutive days to all eligible children in the intervention school. The outcome is the prevalence of parasitemia in the schoolchildren and household members. To assess the impact of the intervention in schoolchildren, 216 children in the intervention school and 216 children in the control school will be randomly selected and assessed at baseline, 1 month and 3 months following the intervention. The same children will be assessed at the 3 school surveys. To assess the impact of the intervention on transmission at the household level, we will enroll 476 household members in the intervention arm and 476 household members in the control arm. Assessments will be conducted at baseline, 1 month and 3 months following the intervention.

ELIGIBILITY:
Inclusion Criteria:

Schools:

1. It is a government-run primary school,
2. Has actively enrolled pupils in primary grades 1-7

School children

1. Are enrolled at the participating school
2. Have parent/guardian consent to receive medication
3. Provided assent for those > 8 years
4. Have no known allergy to study medication (Dihydroartemisinin piperaquine [DP])

Households

1. Have an adult > 18 years of age
2. Agreement of the household head/designate to provide informed consent to participate in the three household surveys (baseline, 1-month post-intervention, and 3-months post-intervention)

Household members

1. Usual resident and present in the household the night before the survey
2. Agreement of resident or parent/guardian to provide informed consent
3. Agreement of children aged 8-17 years to provide assent

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-06-03 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Parasite prevalence | 1 month after the intervention
  Parasitemia measured by microscopy
Parasite prevalence | 3 months after the intervention
  Parasitemia measured by microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere College of Health Sciences, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamya MR, Bakyaita NN, Talisuna AO, Were WM, Staedke SG. Increasing antimalarial drug resistance in Uganda and revision of the national drug policy. Trop Med Int Health. 2002 Dec;7(12):1031-41. doi: 10.1046/j.1365-3156.2002.00974.x. PMID 12460394
- [Background] Yeka A, Nankabirwa J, Mpimbaza A, Kigozi R, Arinaitwe E, Drakeley C, Greenhouse B, Kamya MR, Dorsey G, Staedke SG. Factors associated with malaria parasitemia, anemia and serological responses in a spectrum of epidemiological settings in Uganda. PLoS One. 2015 Mar 13;10(3):e0118901. doi: 10.1371/journal.pone.0118901. eCollection 2015. PMID 25768015
- [Background] Drakeley C, Sutherland C, Bousema JT, Sauerwein RW, Targett GA. The epidemiology of Plasmodium falciparum gametocytes: weapons of mass dispersion. Trends Parasitol. 2006 Sep;22(9):424-30. doi: 10.1016/j.pt.2006.07.001. Epub 2006 Jul 17. PMID 16846756
- [Background] Nankabirwa J, Wandera B, Kiwanuka N, Staedke SG, Kamya MR, Brooker SJ. Asymptomatic Plasmodium infection and cognition among primary schoolchildren in a high malaria transmission setting in Uganda. Am J Trop Med Hyg. 2013 Jun;88(6):1102-1108. doi: 10.4269/ajtmh.12-0633. Epub 2013 Apr 15. PMID 23589533
- [Background] Nankabirwa J, Brooker SJ, Clarke SE, Fernando D, Gitonga CW, Schellenberg D, Greenwood B. Malaria in school-age children in Africa: an increasingly important challenge. Trop Med Int Health. 2014 Nov;19(11):1294-309. doi: 10.1111/tmi.12374. Epub 2014 Aug 22. PMID 25145389
- [Background] Nankabirwa J, Cundill B, Clarke S, Kabatereine N, Rosenthal PJ, Dorsey G, Brooker S, Staedke SG. Efficacy, safety, and tolerability of three regimens for prevention of malaria: a randomized, placebo-controlled trial in Ugandan schoolchildren. PLoS One. 2010 Oct 19;5(10):e13438. doi: 10.1371/journal.pone.0013438. PMID 20976051
- [Background] Nankabirwa JI, Wandera B, Amuge P, Kiwanuka N, Dorsey G, Rosenthal PJ, Brooker SJ, Staedke SG, Kamya MR. Impact of intermittent preventive treatment with dihydroartemisinin-piperaquine on malaria in Ugandan schoolchildren: a randomized, placebo-controlled trial. Clin Infect Dis. 2014 May;58(10):1404-12. doi: 10.1093/cid/ciu150. Epub 2014 Mar 12. PMID 24621953